CLINICAL TRIAL: NCT06691503
Title: A Phase II Clinical Trial of Mediastinoscopic-assisted Transhiatal Laparoscopic Esophagectomy for Early-stage Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: A Clinical Trial of Esophagectomy for Esophageal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Weijie Ye, Investigator, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL-5010-2019-03-02
Record Dates: First submitted 2024-11-08; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Intervention Model Description: Single Group:mediastinoscopic-assisted transhiatal laparoscopic esophagectomy (MATLE);Thirty-five eligible patients with ESCC were assigned to the MATLE group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mediastinoscopic-assisted transhiatal laparoscopic esophagectomy (MATLE) (Experimental)
  Interventions: Procedure: mediastinoscopic-assisted transhiatal laparoscopic esophagectomy (MATLE)

INTERVENTIONS:
Procedure: mediastinoscopic-assisted transhiatal laparoscopic esophagectomy (MATLE) — mediastinoscopic-assisted transhiatal laparoscopic esophagectomy (MATLE)

SUMMARY:
Brief Summary The pathological type of esophageal cancer (EC) in most patients in East Asia is esophageal squamous cell carcinoma (ESCC). Surgery is the primary treatment for EC. This study compared the feasibility and safety of mediastinoscopic-assisted transhiatal laparoscopic esophagectomy (MATLE) with video-assisted thoracoscopic esophagectomy (VATE).

Thirty-five eligible patients with ESCC were assigned to the MATLE group, while seventy matched patients were assigned to the VATE group. The study compared perioperative outcomes and lymph node dissection between the two groups. Additionally, the Kaplan-Meier method was employed to estimate Disease-Free Survival (DFS) and Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* previously untreated
* histologically confirmed
* potentially resectable thoracic ESCC clinically staged as T1b-3N0M0 or Tis-1aN0M0 who was not suitable for endoscopic resection according to the 8th edition of the American Joint Committee on Cancer staging system and National Comprehensive Cancer Network Clinical Practice Guidelines in Esophageal and Esophagogastric Junction Cancers
* age 18-70 years,
* normal hematologic and organ function -Karnofsky Performance Scale (KPS) was assessed as 100 or 90

Exclusion Criteria:

* a history of other malignancies
* severe comorbidities
* active autoimmune disease
* prior non-infectious pneumonitis or interstitial lung disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) and Overall Survival (OS) | DFS : From date of surgery until the date of first documented progression , assessed up to 100 months; OS :From date of surgery until the date of death, assessed up to 100 months
  Disease-free Survival (DFS) was calculated from the date of the operation to the date of tumor recurrence or the last follow-up. Overall Survival (OS) was calculated from the date of the operation to the date of death or the last follow-up. Follow-up was conducted via telephone or outpatient service.

CONTACTS AND LOCATIONS:
Locations (1):
- 651 Dongfeng Road East, Yuexiu District, Guangzhou, P.R. China, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No